CLINICAL TRIAL: NCT05503251
Title: Effect of Early Integrated Neuropsychological Care in Patients With Brain Metastases - A Phase 2 Randomized Controlled Trial
Brief Title: Neuropsychological Care for Maintaining Quality of Life After Radiation Therapy in Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Joshua Palmer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-21074; NCI-2022-02216 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — Practice Guidelines as Topic; Standard of Care; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (neuropsychological evaluation) (Experimental): Patients undergo neuropsychological evaluations with a certified neuropsychologist at baseline, 3 months, and 6 months.
  Interventions: Behavioral: Neuropsychological Assessment; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Behavioral: Neuropsychological Assessment — Undergo neuropsychological evaluation
  Other Names: Neuropsychological Examination
  Arms: Arm I (neuropsychological evaluation)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of neuropsychological evaluation and intervention in maintaining quality of life after radiation therapy in patients with cancer that has spread to the brain (metastases). Quality of life refers to the overall enjoyment of life. It holds varying meanings for different people and may evolve over time. For some individuals it implies autonomy, empowerment, capability, and choice; for others, security, social integration, or freedom from stress or illness. Neuropsychological evaluation is used to examine the cognitive (thinking) consequences of brain damage, brain disease, and severe mental illness. Deterioration of both quality of life and cognitive function is common when receiving radiation to the brain. Neuropsychological evaluation with a certified neuropsychologist may improve quality of life or cognitive function after radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of neuropsychological assessment and follow up on preventing decline of quality of life (QOL) as evaluated by the Functional Assessment of Cancer Therapy Scale-Brain (FACT-Br) score (validated QOL tool for brain metastases).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of early neuropsychological assessment and neurocognitive rehabilitation by a neuropsychologist on prevention of neurocognitive decline in patients treated with radiation to brain metastases as evaluated by the Hopkins Verbal Learning Test-Revised (HVLT-R) Delay Recall, Trail Making Test A/B (TMT A/B), and Controlled Oral Word Association Test (COWAT), and Patient Reported Outcomes Measurement Information System (PROMIS)-8 assessment.

II. To identify subsets of patients treated with whole brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) who receive greater benefits of neuropsychologic evaluation through examining baseline Fact-Br, HVLT-R, TMT A/B, COWAT, and PROMIS-8 completed prior to radiation therapy delivery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo neuropsychological evaluations with a certified neuropsychologist at baseline, 3 months, and 6 months.

ARM II: Patients receive usual care.

After completion of standard of care radiation therapy, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV histologic diagnosis of solid tumor
* Patient will be treated with radiation therapy for brain metastases
* Primarily English-speaking patient
* Graded Prognostic Assessment (GPA) >= 2 (estimated survival > 6 months)

Exclusion Criteria:

* Patient received prior whole brain radiation therapy to the brain
* Patient has multiple sclerosis, Alzheimer's, dementia, or mental disability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) | Up to 12 months after radiation therapy
  Will be measured by the Functional Assessment of Cancer Therapy Scale-Brain instrument. Linear models will be employed to measure QOL score (converted to a 0- to 100-point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Palmer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu